CLINICAL TRIAL: NCT05801653
Title: Health Effects of Oat and Oat Bioactives in Human
Brief Title: Health Effects of Oat Bioactives (Betaglucan) in Human
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Swedish Foundation for Strategic Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Dnr. 2018/658 (del 4)
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oat meal 1 (Experimental): The test portion is based on 30 gram available carbohydrates with added x amount oat betaglucan. Test portion consumed as a breakfast meal prior to determinations of test variables in the morning
  Interventions: Dietary Supplement: Effects of Oat and Oat Components on Cardiometabolic risk variables
- Oat meal 2 (Experimental): The test portion is based on 30 gram available carbohydrates with added y amount of oat betaglucan. Test portion consumed as a breakfast meal prior to determinations of test variables in the morning
  Interventions: Dietary Supplement: Effects of Oat and Oat Components on Cardiometabolic risk variables
- Oat meal 3 (Experimental): The test portion is based on 30 gram available carbohydrates with added z amount of oat betaglucan. Test portion consumed as a breakfast meal prior to determinations of test variables in the morning
  Interventions: Dietary Supplement: Effects of Oat and Oat Components on Cardiometabolic risk variables
- Reference (Placebo Comparator): The test portion is based on 30 gram available carbohydrates without added oat betaglucan. Test portion consumed as a breakfast meal prior to determinations of test variables in the morning
  Interventions: Dietary Supplement: Effects of Oat and Oat Components on Cardiometabolic risk variables

INTERVENTIONS:
Dietary Supplement: Effects of Oat and Oat Components on Cardiometabolic risk variables — Oat and oat bioactive components consumed as breakfast meal.

SUMMARY:
Aim of the study is to investigate health effects of oats and oat derived components, in human intervention studies, with the purpose to build new knowledge for development of cardiometabolic protective foods.

DETAILED DESCRIPTION:
The overall goal is to increase the knowledge which can be used for the development of food products with anti-diabetic properties, with the purpose to facilitate healthier food choices for people. More specifically the primary purpose of this project is to evaluate effects in healthy humans on cardiometabolic test markers of oat and oat based product. The new knowledge will form a base for the development of oat based food products with added health values.

ELIGIBILITY:
Inclusion Criteria:

- Healthy adults BMI 18.5 - 28 Kg/m2 Non smokers Consuming a non-vegetarian diet that follows the Nordic diet recommendation.

Exclusion Criteria:

- Fasting blood glucose concentration >6.1 mmol/l Known cardio-metabolic disease (e.g. diabetes, hypertension, metabolic syndrome).

Gastro-intestinal disorders such as IBS (irritable bowel syndrome) that can interfere with the study results, food allergies.

No antibiotics or probiotics should have been consumed within 4 weeks prior to and during the study.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Blood glucose regulation | Time Frame: 0 - 5.5 hours ( at fasting and then repeatedly after breakfast and Standardize lunch)
  Postprandial blood glucose regulation (incremental area under the curve) acute after intake of the test products and at forthcoming meals within 5.5 hours after consumption of test products.

SECONDARY OUTCOMES:
Serum insulin | Time Frame: 0 - 5.5 hours ( at fasting and then repeatedly after breakfast and Standardize lunch)
  Acute effects of postprandial serum insulin concentrations (incremental area under the curve) after intake of the test products.

OTHER OUTCOMES:
Subjective appetite sensations | Time Frame: 0 - 5.5 hours ( at fasting and then repeatedly after breakfast and Standardize lunch)
  Determined with VAS (visual analogue scale) scales (0-100 mm) as a range of subjective sensations related to appetite (such as hunger, desire to eat or fullness)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Nilsson, Principal Investigator — Department of Food Technology, Engineering and Nutrition, Lund Univesity
Locations (1):
- Food Technology, engineering and Nutrition, LTH, Lund University, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No
Raw data